CLINICAL TRIAL: NCT00375596
Title: Study Withdrawn Prior to Determining Official Title
Brief Title: A Study Of The Safety And Effectiveness Of A New Treatment For Allergic Conjunctivitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn without starting or enrolling subjects due to a business decision to not proceed with the project.
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Model: Parallel
Other Study IDs: C-02-06-001
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen; Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ketotifen/vasoconstrictor

SUMMARY:
This study will evaluate the safety and efficacy of a new allergy medication

DETAILED DESCRIPTION:
Study withdrawn prior to determining study details

ELIGIBILITY:
Inclusion Criteria:

* Be at least 6 years of age, of any race, or either gender.
* Have a positive allergic history of ocular allergies and a positive skin test reaction to cat hair/dander, ragweed, tree and/or grass pollen within the past 24 months.
* Have a calculated best-corrected visual acuity of 0.6 logMar or better in each eye as measured using an ETDRS chart.
* Positive bilateral CAC reaction at Visit 1 & 2.

Exclusion Criteria:

* Have any known contraindications, allergies, or sensitivities to the use of any of the study medications, or their components.
* Any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters
* Manifest signs or symptoms of clinically active allergic conjunctivitis in either eye at the baseline slit-lamp exam of any visit

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of a new allergy medication | 0
  STUDY WITHDRAWN PRIOR TO OUTCOME DETERMINATION